CLINICAL TRIAL: NCT00811135
Title: A Single Arm Open-label, Phase II Study of Bevacizumab in Combination With Trastuzumab and Capecitabine as First-line Treatment of Patients With HER2-positive Locally Recurrent or Metastatic Breast Cancer
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Herceptin (Trastuzumab) and Xeloda (Capecitabine) in Patients With HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO21926; 2008-003283-20
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Capecitabine; Trastuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]; Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 15mg/kg iv on day 2 of first 3-week cycle,and on day 1 of subsequent cycles
Drug: capecitabine [Xeloda] — 1000mg/m2 bid po on days 1-14 of each 3-week cycle
Drug: trastuzumab [Herceptin] — 8mg/kg iv loading dose on day 1 of first 3-week cycle, followed by 6mg/kg iv maintenance dose on day 1 of subsequent cycles

SUMMARY:
This single arm study will assess the efficacy and safety of Avastin in combination with Herceptin and Xeloda as first-line treatment of patients with HER2-positive locally recurrent or metastatic breast cancer. Patients will receive 3-weekly treatment cycles of Herceptin (8mg/kg iv on day 1 of first cycle, followed by 6mg/kg iv maintenance dose on day 1 of subsequent cycles), Xeloda (1000mg/m2 bid po on days 1-14 of each treatment cycle) and Avastin (15mg/kg on day 2 of first treatment cycle,and on day 1 of each subsequent cycle).The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* breast cancer with measurable locally recurrent or metastatic lesions;
* candidate for chemotherapy;
* HER2-positive disease;
* ECOG PS of <=2.

Exclusion Criteria:

* previous anticancer therapy for metastatic breast cancer;
* previous radiotherapy for metastatic breast cancer (except for adjuvant radiotherapy >=6 months before enrollment);
* chronic daily treatment with corticosteroids (>=10mg/day), aspirin (>325 mg/day) or clopidogrel (>75mg/day);
* other primary tumor within last 5 years, except for adequately treated cervical cancer in situ, squamous or basal cell skin cancer;
* uncontrolled hypertension or significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (29):
- Denmark (2):
  - Herlev
  - Vejle
- France (12):
  - Aix-en-Provence
  - Béziers
  - Créteil
  - Dechy
  - Lormont
  - Marseille
  - Narbonne
  - Paris
  - Rodez
  - Saint-Jean
  - Saint-Quentin
  - Toulouse
- Russia (2):
  - Moscow
  - Saint Petersburg
- Bratislava, Slovakia
- Spain (8):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Málaga, Malaga
  - Pontevedra, Pontevedra
  - Salamanca, Salamanca
  - Seville, Sevilla
  - Valencia, Valencia
  - Barakaldo, Vizcaya
- Sweden (4):
  - Eskilstuna
  - Sundsvall
  - Uppsala
  - Vaxjo

REFERENCES:
- [Derived] Martin M, Makhson A, Gligorov J, Lichinitser M, Lluch A, Semiglazov V, Scotto N, Mitchell L, Tjulandin S. Phase II study of bevacizumab in combination with trastuzumab and capecitabine as first-line treatment for HER-2-positive locally recurrent or metastatic breast cancer. Oncologist. 2012;17(4):469-75. doi: 10.1634/theoncologist.2011-0344. Epub 2012 Mar 30. PMID 22467666

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening details were taken 28 days prior to baseline. There were 88 participants included from 23 centers.
Groups:
- Trastuzumab + Bevacizumab + Capecitabine: Participants received intravenous (IV) trastuzumab (8 milligrams per kilogram [mg/kg]) for first cycle and then 6 mg/kg for subsequent cycles followed by bevacizumab (15 mg/kg) on Day 1 of each treatment cycles along with capecitabine administered orally to participants at a dose of 1000 milligrams per meter square (mg/m^2) twice daily (BID) on Days 1 to 14 of each treatment cycle until disease progression, unmanageable toxicity or participant request for discontinuation. Treatment cycles were of 3 weeks.
Period: Overall Study
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Started | 88
Completed | 0
Not Completed | 88
Not completed — Adverse Event/Intercurrent Illness | 8
Not completed — Death | 3
Not completed — Protocol Violation | 2
Not completed — Violation of Selection Criteria | 1
Not completed — Refused Treatment | 1
Not completed — Withdrawal by Subject | 3
Not completed — Administrative/Other Unspecified | 11
Not completed — Ongoing | 59

BASELINE CHARACTERISTICS:
Population: The Intention-To-Treat (ITT) population included all participants enrolled in the study who received at least one dose of any study medication.
Groups:
- Trastuzumab + Bevacizumab + Capecitabine: Participants received IV trastuzumab (8 mg/kg) for first cycle and then 6 mg/kg for subsequent cycles followed by bevacizumab (15 mg/kg) on Day 1 of each treatment cycles along with capecitabine administered orally to participants at a dose of 1000 mg/m^2 BID on Days 1 to 14 of each treatment cycle until disease progression, unmanageable toxicity or participant request for discontinuation. Treatment cycles were of 3 weeks.
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Response (BOR) of Confirmed Complete Response (CR) or Partial Response (PR)
Description: Tumor response was assessed using the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.0. BOR was defined as the best response recorded for a participant from the start of treatment until disease progression/recurrence. Percentage of participants with a BOR of confirmed CR or PR (responders) was reported. CR: disappearance of all target and non-target lesions and normalization of tumor marker level; PR: at least a 30 percent (%) decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Confirmed responses were those which were confirmed by a repeat assessment, performed 4 weeks after the criteria for response first met.
Time Frame: Screening until disease progression (assessed at screening, every 6 weeks up to Week 36, thereafter every 9 weeks during treatment period, and then every 3 months during follow-up, up to approximately 4 years)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
percentage of participants | 75.0 [64.6 to 83.6]

2. Secondary Outcome: Number of Participants With Disease Progression or Death
Description: Disease progression was defined as at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
participants | 70

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from enrollment to time of first documented disease progression or death due to any cause, whichever occurred first. Progression: at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. PFS was estimated using Kaplan-Meier methods.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
months | 14.2 [10.5 to 14.9]

4. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: OS was defined as the time from enrollment to death from any cause where enrollment was defined as successfully passed screening visit, enrolled in the study and received first dose of study treatment.
Time Frame: Screening until death (assessed at screening, every 6 weeks up to Week 36, thereafter every 9 weeks during treatment period, and then every 3 months during follow-up, up to approximately 4 years)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
participants | 40

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from enrollment to death from any cause where enrollment was defined as successfully passed screening visit, enrolled in the study and received first dose of study treatment. OS was estimated using Kaplan-Meier methods.
Time Frame: as for outcome 4
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
months | 31.8 [26.3 to 38.2]

6. Secondary Outcome: Number of Participants With Time to Progression (TTP)
Description: TTP was defined as the time from enrollment to first documented disease progression (at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions). TTP was estimated using Kaplan-Meier methods.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
participants | 62

7. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from enrollment to first documented disease progression (at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions).
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
months | 14.5 [11.0 to 17.0]

8. Secondary Outcome: Number of Participants With Response
Description: Participants who had CR or PR were considered as responders. CR: disappearance of all target and non-target lesions and normalization of tumor marker level; PR: at least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
participants | 66

9. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from the first recorded response (CR/PR) to the date of first documented progression or death. CR: disappearance of all target lesions and non-target lesions and normalization of tumor marker level. PR: at least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD. Progression: at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. DR was estimated using Kaplan-Meier methods.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Number analyzed (Participants) | 88
months | 12.7 [10.2 to 17.7]

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last study treatment dose (maximum treatment time = approximately 44 months)
Description: The safety population comprised of all participants who received at least one dose of any study medication.
Arm/Group | Trastuzumab + Bevacizumab + Capecitabine
Serious Adverse Events (participants affected / at risk) | 20/88
Other Adverse Events (participants affected / at risk) | 81/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Bevacizumab + Capecitabine (N=88)
Cardiac Failure (Cardiac disorders) | 2
Intracardiac thrombus (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 1
Erysipelas (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Bevacizumab + Capecitabine (N=88)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 65
Nail disorder (Skin and subcutaneous tissue disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 37
Nausea (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 15
Stomatitis (Gastrointestinal disorders) | 10
Abdominal pain upper (Gastrointestinal disorders) | 9
Gingival bleeding (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 5
Haemorrhoids (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 32
Pyrexia (General disorders) | 18
Fatigue (General disorders) | 11
Mucosal inflammation (General disorders) | 10
Oedema peripheral (General disorders) | 6
Chest pain (General disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Hypertension (Vascular disorders) | 34
Headache (Nervous system disorders) | 14
Proteinuria (Renal and urinary disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 12
Urinary tract infection (Infections and infestations) | 7
Respiratory tract infection viral (Infections and infestations) | 5
Weight decreased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.